CLINICAL TRIAL: NCT01887093
Title: The Influence of Regular Walking at Different Times of Day on Blood Lipids and Inflammatory Markers in Sedentary Patients With Coronary Artery Disease
Brief Title: The Influence of Walking at Different Times of Day on Blood Lipids and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiao-Qing Lian, The First Hospital of Nanjing Medical University, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NSFC(No. 81270255); 81270255 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2013-06-22; First posted 2013-06-26 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; walking; lipids; inflammatory markers; time of day
MeSH Terms: conditions — Coronary Artery Disease | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Morning walking (Experimental): Participants were requested to walk in the morning at the speed of 2.5 miles/h for 30 min/day or more on at least 5 days/week for a period of 12 weeks. We demanded everyone to record the situation of walking including duration, distance and time daily in a log book. Each participant was telephoned at least once a week to ensure the adherence to the exercise program. Patients were called back every month to hand in the log book and to understand the information about medication use. Furthermore, at the beginning and end of the 12-week program, both the walking groups were supervised by researchers to walk for continuous three days and the duration and distance of walking were recorded.
  Interventions: Behavioral: walking
- Evening walking (Experimental): Participants were requested to walk in the evening at the speed of 2.5 miles/h for 30 min/day or more on at least 5 days/week for a period of 12 weeks. We demanded everyone to record the situation of walking including duration, distance and time daily in a log book. Each participant was telephoned at least once a week to ensure the adherence to the exercise program. Patients were called back every month to hand in the log book and to understand the information about medication use. Furthermore, at the beginning and end of the 12-week program, both the walking groups were supervised by researchers to walk for continuous three days and the duration and distance of walking were recorded.
  Interventions: Behavioral: walking
- No walking (No Intervention): The control group was requested to maintain their usual level of physical activity.

INTERVENTIONS:
Behavioral: walking — Participants in both walking groups were requested to walk at the speed of 2.5 miles/h for 30 min/day or more on at least 5 days/week for a period of 12 weeks.One group was asked to walk in the morning and the other group was asked to walk in the evening.
  Arms: Evening walking; Morning walking

SUMMARY:
It has been well known that moderate and regular levels of physical activity has a favorable effect on many of the established risk factors related to coronary artery disease (CAD). Given that exercise in the morning has a greater potential for inducing sudden cardiac death and myocardial ischemia, it may be sensible for patients with CAD not to take exercise at this time. Our previous study indicated that the protective effect of exercise in the evening was greater than morning. However, which times of day to exercise could achieve the greatest improvements in lipids and inflammatory markers remains unclear. The purpose of the present study was to investigate the responses of lipid profiles and inflammatory markers to walking at different times of day in sedentary patients with CAD.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 330 patients with CAD between the ages of 40 and 80 years were recruited from the inpatient cardiology department of the First Affiliated Hospital of Nanjing Medical University. Informed consent was obtained from each participant after explaining the study protocols. Patients were randomly assigned to one of the three groups: control group (n=110), morning walking group (n=110) or evening walking group (n=110). The control group was requested to maintain their usual level of physical activity. Participants in both walking groups were requested to walk at the speed of 2.5 miles/h for 30 min/day or more on at least 5 days/week for a period of 12 weeks. The protocol of exercise was identical, while the difference between the two groups was that one group was asked for walking in the morning and the other group walking in the evening. Each participant was telephoned at least once a week to ensure the adherence to the exercise program. Patients were called back every month to understand the information about walking and medication use. In the intervention groups, subjects whose compliance rate with their respectively walking program were less than 85% were excluded in the analysis. Additionally, all the participants were given an advice on quitting smoking and were provided with similar diets by a nutritionist, as to caloric intake and nutrients. Total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, lipoprotein a, white blood cell count and platelet count, fibrinogen were measured before and after the intervention.

The Kolmogorov-Smirnov test was used to check the normal distribution of all continuous variables. The values of normal distribution were expressed as mean±SD, and non-normal distribution data were presented as median (interquartile range). Baseline differences between groups were determined by one-way analysis of variance and chi-square analyses. Baseline and follow-up values within each group were compared using the paired t test. General linear models were used to adjust the differences in baseline values for dependent variables. And two-way ANOVA was used for determination of the improvements of lipids and inflammatory markers in three groups. The significance level was defined as P<0.05. All analyses were carried out using SPSS version 13.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were younger than 80 years;
2. They had been diagnosed with coronary artery disease by coronary angiography (at least 1 main coronary artery having >50% luminal diameter stenosis);
3. They were able to walk but had a sedentary lifestyle which was defined as no regular physical activity in excess of 30 min/day, for more than 3 days/week over the last 3 months.

Exclusion Criteria:

1. valvular heart disease;
2. atrial fibrillation;
3. cardiomyopathy;
4. myocarditis;
5. uncontrolled chronic diseases;
6. congestive heart failure or ejection fraction <50% by echocardiogram.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Blood lipids and inflammatory markers | 12 weeks
  Blood lipids include total cholesterol, triglycerides, high-density lipoprotein cholesterol,low-density lipoprotein cholesterol, lipoprotein a;inflammatory markers include white blood cell count, platelet count, fibrinogen

SECONDARY OUTCOMES:
Blood lipids and inflammatory markers | 24 weeks
  Blood lipids include total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein, lipoprotein a; inflammatory markers include white blood cell count, platelet count, fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Qing Lian, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Cardiology, the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Boardley D, Fahlman M, Topp R, Morgan AL, McNevin N. The impact of exercise training on blood lipids in older adults. Am J Geriatr Cardiol. 2007 Jan-Feb;16(1):30-5. doi: 10.1111/j.1076-7460.2007.05353.x. PMID 17215640
- [Background] Ainsworth BE, Haskell WL, Whitt MC, Irwin ML, Swartz AM, Strath SJ, O'Brien WL, Bassett DR Jr, Schmitz KH, Emplaincourt PO, Jacobs DR Jr, Leon AS. Compendium of physical activities: an update of activity codes and MET intensities. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S498-504. doi: 10.1097/00005768-200009001-00009. PMID 10993420
- [Background] Andreotti F, Davies GJ, Hackett DR, Khan MI, De Bart AC, Aber VR, Maseri A, Kluft C. Major circadian fluctuations in fibrinolytic factors and possible relevance to time of onset of myocardial infarction, sudden cardiac death and stroke. Am J Cardiol. 1988 Sep 15;62(9):635-7. doi: 10.1016/0002-9149(88)90669-8. No abstract available. PMID 3137799
- [Background] Elherik K, Khan F, McLaren M, Kennedy G, Belch JJ. Circadian variation in vascular tone and endothelial cell function in normal males. Clin Sci (Lond). 2002 May;102(5):547-52. PMID 11980574
- [Background] Fahlman MM, Boardley D, Lambert CP, Flynn MG. Effects of endurance training and resistance training on plasma lipoprotein profiles in elderly women. J Gerontol A Biol Sci Med Sci. 2002 Feb;57(2):B54-60. doi: 10.1093/gerona/57.2.b54. PMID 11818424
- [Background] Geffken DF, Cushman M, Burke GL, Polak JF, Sakkinen PA, Tracy RP. Association between physical activity and markers of inflammation in a healthy elderly population. Am J Epidemiol. 2001 Feb 1;153(3):242-50. doi: 10.1093/aje/153.3.242. PMID 11157411
- [Background] Jahangard T, Torkaman G, Ghoosheh B, Hedayati M, Dibaj A. The effect of short-term aerobic training on coagulation and fibrinolytic factors in sedentary healthy postmenopausal women. Maturitas. 2009 Dec 20;64(4):223-7. doi: 10.1016/j.maturitas.2009.09.003. Epub 2009 Oct 24. PMID 19854593
- [Background] Jones H, Pritchard C, George K, Edwards B, Atkinson G. The acute post-exercise response of blood pressure varies with time of day. Eur J Appl Physiol. 2008 Oct;104(3):481-9. doi: 10.1007/s00421-008-0797-4. Epub 2008 Jun 20. PMID 18566827
- [Background] Kanaley JA, Weltman JY, Pieper KS, Weltman A, Hartman ML. Cortisol and growth hormone responses to exercise at different times of day. J Clin Endocrinol Metab. 2001 Jun;86(6):2881-9. doi: 10.1210/jcem.86.6.7566. PMID 11397904
- [Background] Kelley GA, Kelley KS, Tran ZV. Walking, lipids, and lipoproteins: a meta-analysis of randomized controlled trials. Prev Med. 2004 May;38(5):651-61. doi: 10.1016/j.ypmed.2003.12.012. PMID 15066369
- [Background] Kraus WE, Houmard JA, Duscha BD, Knetzger KJ, Wharton MB, McCartney JS, Bales CW, Henes S, Samsa GP, Otvos JD, Kulkarni KR, Slentz CA. Effects of the amount and intensity of exercise on plasma lipoproteins. N Engl J Med. 2002 Nov 7;347(19):1483-92. doi: 10.1056/NEJMoa020194. PMID 12421890
- [Background] Lee CD, Folsom AR, Nieto FJ, Chambless LE, Shahar E, Wolfe DA. White blood cell count and incidence of coronary heart disease and ischemic stroke and mortality from cardiovascular disease in African-American and White men and women: atherosclerosis risk in communities study. Am J Epidemiol. 2001 Oct 15;154(8):758-64. doi: 10.1093/aje/154.8.758. PMID 11590089
- [Background] Lippi G, Franchini M, Salvagno GL, Montagnana M, Guidi GC. Higher morning serum cortisol level predicts increased fibrinogen but not shortened APTT. J Thromb Thrombolysis. 2008 Oct;26(2):103-5. doi: 10.1007/s11239-007-0074-0. Epub 2007 Jul 13. PMID 17629773
- [Background] Maresca G, Di Blasio A, Marchioli R, Di Minno G. Measuring plasma fibrinogen to predict stroke and myocardial infarction: an update. Arterioscler Thromb Vasc Biol. 1999 Jun;19(6):1368-77. doi: 10.1161/01.atv.19.6.1368. PMID 10364066
- [Derived] Lian XQ, Zhao D, Zhu M, Wang ZM, Gao W, Zhao H, Zhang DG, Yang ZJ, Wang LS. The influence of regular walking at different times of day on blood lipids and inflammatory markers in sedentary patients with coronary artery disease. Prev Med. 2014 Jan;58:64-9. doi: 10.1016/j.ypmed.2013.10.020. Epub 2013 Nov 4. PMID 24201089